CLINICAL TRIAL: NCT00016991
Title: A Phase II Study of ZD 1839 (NSC 715055) for Patients With First Relapse Glioblastoma Multiforme
Brief Title: ZD 1839 in Treating Patients With Glioblastoma Multiforme in First Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Henry Friedman, MD, Duke UMC
Purpose: Treatment
Other Study IDs: 2421; DUMC-2421-03-2R2; DUMC-2421-01-2; NCI-1253; CDR0000068639 (Other: NCI)
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Gefitinib

INTERVENTIONS:
Drug: gefitinib

SUMMARY:
RATIONALE: Biological therapies such as ZD 1839 may interfere with the growth of tumor cells and slow the growth of glioblastoma multiforme.

PURPOSE: Phase II trial to study the effectiveness of ZD 1839 in treating patients who have glioblastoma multiforme in first relapse.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of ZD 1839 in patients with glioblastoma multiforme in first relapse.
* Determine the pharmacokinetics and toxicity of this drug in these patients.
* Assess the relationship between epidermal growth factor receptor status in these patients and activity of this drug.

OUTLINE: Patients receive oral ZD 1839 once daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for at least 6 months.

PROJECTED ACCRUAL: A total of 53 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme in first relapse

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal:

* Creatinine less than 1.5 times ULN

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No prior allergic reactions to compounds of similar chemical or biologic composition to ZD 1839
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Ocular inflammation must be fully treated before study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* Must be on stable dose of steroids for at least 1 week

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* At least 1 week since prior surgery

Other:

* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV
* No concurrent enzyme-inducing anticonvulsant drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States